CLINICAL TRIAL: NCT06346769
Title: Clinical Evaluation of Composite Restorations Performed by Placing Polyethylene Fiber in Endodontically Treated Posterior Teeth
Brief Title: Composite Restorations Performed by Placing Polyethylene Fiber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Merve Gurses, Assistant Proffesor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SelcukB
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Endodontically Treated Teeth
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 'O' shape polyethylene fiber (Experimental)
  Interventions: Other: Polyethylene Fiber
- mesiodistal I shape polyethylene fiber (Experimental)
  Interventions: Other: Polyethylene Fiber
- buccolingual I shape polyethylene fiber (Experimental)
  Interventions: Other: Polyethylene Fiber

INTERVENTIONS:
Other: Polyethylene Fiber — In the restoration of the endodontically treated posterior teeth, polyethylene fiber was placed in different directions ('O' shape, mesiodistal I shape, buccolingual I shape) according to the amount of remaining tooth tissue and cavity preparation.

SUMMARY:
This study aimed to evaluate the 12-month clinical performance of direct composite restorations by placing polyethylene fibers in different directions in endodontically treated posterior teeth. In this clinical study, Clearfil SE Bond (Kuraray/Japan) adhesive system, G-aenial Universal Injectable (GC/Tokyo, Japan), G-aenial A'chord (GC/Tokyo, Japan) composites, and polyethylene fiber (Ribbond, USA) were used. In the restoration of the teeth included in the study, polyethylene fiber was placed in different directions according to the amount of remaining tooth tissue and cavity preparation. The restorations were divided into three groups according to the direction of fiber placement ('O' shape, mesiodistal I shape, buccolingual I shape) (n=12). Restorations were evaluated according to modified USPHS criteria in 1st week and 6th months from the placement date. The Chi-square test was used for statistical analysis of the difference between the groups, and the Cochran Q test was used for the significance of the difference between time-dependent changes within each group (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

A patient presenting with;

1. over 18 years of age
2. a normal periodontal status and good general health
3. endodontically treated premolar and molar teeth
4. teeth in contact with the opposing tooth and subjected to normal occlusal forces
5. attend follow-up appointments

Exclusion Criteria:

1. poor oral hygiene status
2. those with severe or chronic periodontitis
3. absence of adjacent and antagonist teeth
4. potential behavioral problems (e.g. bruxism)
5. allergy to any product used in the study
6. systemically unhealthy
7. pregnant and lactating women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Retention | Seventh day, sixth month, twelfth month
  No loss of restorative material
Color match | Seventh day, sixth month, twelfth month
  The restoration matches the adjacent tooth structure in color and translucency
Marginal Discoloration | Seventh day, sixth month, twelfth month
  There is no discoloration anywhere on the margin between the restoration and the tooth structure
Marginal adaptation | Seventh day, sixth month, twelfth month
  There is no visible evidence of a crevice along the margin into which the explorer will penetrate
Secondary caries | Seventh day, sixth month, twelfth month
  No evidence of secondary caries
Surface texture | Seventh day, sixth month, twelfth month
  The surface of the restoration does not have any defects
Anatomical form | Seventh day, sixth month, twelfth month
  The restoration is continuous with the existing anatomic form

CONTACTS AND LOCATIONS:
Overall Officials: MERVE GÜRSES, Principal Investigator — Selcuk University, Faculty of Dentistry
Locations (2):
- Turkey (Türkiye) (2):
  - Selcuk University, Faculty of Dentistry, Restorative Dentistry Department, Konya
  - Selcuk University, Faculty of Dentistry, Konya

IPD SHARING:
Plan to Share IPD: No